CLINICAL TRIAL: NCT04083859
Title: A Pragmatic Randomized-Controlled Trial of a Digital Outreach Intervention for Lung Cancer Screening: mPATH-Lung (Mobile Patient Technology for Health-Lung)
Brief Title: Digital Outreach Intervention for Lung Cancer Screening
Acronym: mPATH-Lung
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: IRB00060382; IRB00060382 (Other: Institutional Review Board - Wake Forest University Health Science); 1R01CA237240 (NIH)
Record Dates: First submitted 2019-08-30; First posted 2019-09-10 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer
Keywords: Mass screening; Early detection of cancer; Digital health interventions; Decision making, computer assisted
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mPATH-Lung (Experimental): Participants randomized to the mPATH arm will be shown a 5-minute animated LCS decision aid video, personalized risk/benefit information, and a values clarification exercise. The participants in this group will be given an option to request a screening appointment via the program.
  Interventions: Other: mPATH-Lung
- Usual care (CONTROL) (Placebo Comparator): Participants randomized to the control arm will be advised that they qualified for lung cancer screening and directed to speak with their provider if interested. The web app then displayed a 5-minute video about exercise for lung health before ending. They will not be offered the opportunity to estimate their predicted benefits and harms of screening or to request a lung cancer screening visit.
  Interventions: Other: Lung health video

INTERVENTIONS:
Other: mPATH-Lung — A web-based program that determines patients eligibility for lung cancer screening (LCS), informs them of LCS, presents them with personalized risk-benefit information, helps them make a screening decision, and helps them schedule a LCS clinic appointment.
  Arms: mPATH-Lung
Other: Lung health video — Web-based video about guideline recommended exercise for lung health
  Arms: Usual care (CONTROL)

SUMMARY:
mPATH-Lung (mobile Patient Technology for Health - Lung) is an innovative digital outreach program that identifies patients who qualify for lung cancer screening and helps them get screened. The study will: 1) Determine the effect of mPATH-Lung on receipt of lung cancer screening in a pragmatic randomized-controlled trial conducted with primary care patients in two large health networks, 2) Elucidate the drivers of patients' screening decisions and screening behavior; and 3) Explore implementation outcomes that will impact the sustainability and dissemination of mPATH-Lung using program data, surveys, and interviews.

This project will determine how mPATH-Lung affects patients' screening decisions and their completion of screening.

DETAILED DESCRIPTION:
Primary Objective: Determine the effectiveness of mPATH-Lung on receipt of LCS in a randomized pragmatic clinical trial of 1318 patients recruited from two large health networks, Wake Forest Baptist Health and the University of North Carolina at Chapel Hill.

Secondary Objectives:

* Elucidate the drivers of patients' decisions to receive or forgo LCS through a values clarification exercise embedded within mPATH-Lung and supplemental semi-structured interviews of at least 50 patients.
* Assess several critical implementation outcomes (reach, acceptability, and appropriateness) to inform the sustainability and scalability of mPATH-Lung across diverse primary care settings

ELIGIBILITY:
Inclusion Criteria:

* Meet the Medicare criteria for lung cancer screening, as updated in February 2022:

  * Age 50 - 77 years
  * Smoked at least 20 pack years
  * Current smoker or quit smoking within the past 15 years
* Be scheduled to see a primary care provider within the health network in the next 3-4 weeks
* Have a patient portal account or cellphone number listed in the electronic health record

Exclusion Criteria:

* Patients flagged as needing a language interpreter in the electronic health record (electronic messages and intervention is delivered in English only).
* Those for whom lung cancer screening would be inappropriate:

  * Prior history of lung cancer
  * Chest CT within the last 12 months
  * Those with medical conditions predicting shorter life expectancy
  * Patients whose home address is not within the state of North Carolina. (Due to telehealth guidelines)

Ages: 50 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26998 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P Miller, MD, MS, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - University of North Carolina- Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified individual participant data that underlie our published or presented results with researchers who provide a methodologically sound proposal. Use of the data will be limited to achieve the aims in their submitted proposal. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol
Time Frame: We will make the de-identified data available within one year of the publication of the relevant results. Data will remain available for at least 5 years from the last publication of results.
Access Criteria: Researchers desiring data access must provide a methodologically sound proposal to the study principal investigator. Use of the data will be limited to achieve the aims in their submitted proposal. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Viale PH. The American Cancer Society's Facts & Figures: 2020 Edition. J Adv Pract Oncol. 2020 Mar;11(2):135-136. doi: 10.6004/jadpro.2020.11.2.1. Epub 2020 Mar 1. No abstract available. PMID 33532112
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] Pinsky PF, Church TR, Izmirlian G, Kramer BS. The National Lung Screening Trial: results stratified by demographics, smoking history, and lung cancer histology. Cancer. 2013 Nov 15;119(22):3976-83. doi: 10.1002/cncr.28326. Epub 2013 Aug 26. PMID 24037918
- [Background] Moyer VA; U.S. Preventive Services Task Force. Screening for lung cancer: U.S. Preventive Services Task Force recommendation statement. Ann Intern Med. 2014 Mar 4;160(5):330-8. doi: 10.7326/M13-2771. PMID 24378917
- [Background] Wender R, Fontham ET, Barrera E Jr, Colditz GA, Church TR, Ettinger DS, Etzioni R, Flowers CR, Gazelle GS, Kelsey DK, LaMonte SJ, Michaelson JS, Oeffinger KC, Shih YC, Sullivan DC, Travis W, Walter L, Wolf AM, Brawley OW, Smith RA. American Cancer Society lung cancer screening guidelines. CA Cancer J Clin. 2013 Mar-Apr;63(2):107-17. doi: 10.3322/caac.21172. Epub 2013 Jan 11. PMID 23315954
- [Background] Jaklitsch MT, Jacobson FL, Austin JH, Field JK, Jett JR, Keshavjee S, MacMahon H, Mulshine JL, Munden RF, Salgia R, Strauss GM, Swanson SJ, Travis WD, Sugarbaker DJ. The American Association for Thoracic Surgery guidelines for lung cancer screening using low-dose computed tomography scans for lung cancer survivors and other high-risk groups. J Thorac Cardiovasc Surg. 2012 Jul;144(1):33-8. doi: 10.1016/j.jtcvs.2012.05.060. PMID 22710039
- [Background] Centers for Medicare & Medicaid Services. Final National Coverage Determination on Screening for Lung Cancer with Low Dose Computed Tomography (LDCT) (CAG-00439N).; 2015. https://www.cms.gov/medicare-coverage-database/details/nca-decision-memo.aspx?NCAId=274. Accessed November 10, 2015.
- [Background] Jemal A, Fedewa SA. Lung Cancer Screening With Low-Dose Computed Tomography in the United States-2010 to 2015. JAMA Oncol. 2017 Sep 1;3(9):1278-1281. doi: 10.1001/jamaoncol.2016.6416. PMID 28152136
- [Background] Bach PB, Mirkin JN, Oliver TK, Azzoli CG, Berry DA, Brawley OW, Byers T, Colditz GA, Gould MK, Jett JR, Sabichi AL, Smith-Bindman R, Wood DE, Qaseem A, Detterbeck FC. Benefits and harms of CT screening for lung cancer: a systematic review. JAMA. 2012 Jun 13;307(22):2418-29. doi: 10.1001/jama.2012.5521. PMID 22610500
- [Background] Harris RP, Sheridan SL, Lewis CL, Barclay C, Vu MB, Kistler CE, Golin CE, DeFrank JT, Brewer NT. The harms of screening: a proposed taxonomy and application to lung cancer screening. JAMA Intern Med. 2014 Feb 1;174(2):281-5. doi: 10.1001/jamainternmed.2013.12745. PMID 24322781
- [Background] Veronesi G, Maisonneuve P, Bellomi M, Rampinelli C, Durli I, Bertolotti R, Spaggiari L. Estimating overdiagnosis in low-dose computed tomography screening for lung cancer: a cohort study. Ann Intern Med. 2012 Dec 4;157(11):776-84. doi: 10.7326/0003-4819-157-11-201212040-00005. PMID 23208167
- [Background] Patz EF Jr. Lung cancer screening, overdiagnosis bias, and reevaluation of the Mayo Lung Project. J Natl Cancer Inst. 2006 Jun 7;98(11):724-5. doi: 10.1093/jnci/djj226. No abstract available. PMID 16757691
- [Background] Kovalchik SA, Tammemagi M, Berg CD, Caporaso NE, Riley TL, Korch M, Silvestri GA, Chaturvedi AK, Katki HA. Targeting of low-dose CT screening according to the risk of lung-cancer death. N Engl J Med. 2013 Jul 18;369(3):245-254. doi: 10.1056/NEJMoa1301851. PMID 23863051
- [Background] Brenner A, Howard K, Lewis C, Sheridan S, Crutchfield T, Hawley S, Reuland D, Kistler C, Pignone M. Comparing 3 values clarification methods for colorectal cancer screening decision-making: a randomized trial in the US and Australia. J Gen Intern Med. 2014 Mar;29(3):507-13. doi: 10.1007/s11606-013-2701-0. Epub 2013 Nov 23. PMID 24272830
- [Background] Reuland DS, Cubillos L, Brenner AT, Harris RP, Minish B, Pignone MP. A pre-post study testing a lung cancer screening decision aid in primary care. BMC Med Inform Decis Mak. 2018 Jan 12;18(1):5. doi: 10.1186/s12911-018-0582-1. PMID 29325548
- [Background] Fagerlin A, Pignone M, Abhyankar P, Col N, Feldman-Stewart D, Gavaruzzi T, Kryworuchko J, Levin CA, Pieterse AH, Reyna V, Stiggelbout A, Scherer LD, Wills C, Witteman HO. Clarifying values: an updated review. BMC Med Inform Decis Mak. 2013;13 Suppl 2(Suppl 2):S8. doi: 10.1186/1472-6947-13-S2-S8. Epub 2013 Nov 29. PMID 24625261
- [Background] Elwyn G, O'Connor A, Stacey D, Volk R, Edwards A, Coulter A, Thomson R, Barratt A, Barry M, Bernstein S, Butow P, Clarke A, Entwistle V, Feldman-Stewart D, Holmes-Rovner M, Llewellyn-Thomas H, Moumjid N, Mulley A, Ruland C, Sepucha K, Sykes A, Whelan T; International Patient Decision Aids Standards (IPDAS) Collaboration. Developing a quality criteria framework for patient decision aids: online international Delphi consensus process. BMJ. 2006 Aug 26;333(7565):417. doi: 10.1136/bmj.38926.629329.AE. Epub 2006 Aug 14. PMID 16908462
- [Background] Edwards A, Elwyn G. Shared Decision-Making in Health Care: Achieving Evidence-Based Patient Choice. Oxford: Oxford University Press; 2009.
- [Background] Carter-Harris L, Brandzel S, Wernli KJ, Roth JA, Buist DSM. A qualitative study exploring why individuals opt out of lung cancer screening. Fam Pract. 2017 Apr 1;34(2):239-244. doi: 10.1093/fampra/cmw146. PMID 28122849
- [Background] Ali N, Lifford KJ, Carter B, McRonald F, Yadegarfar G, Baldwin DR, Weller D, Hansell DM, Duffy SW, Field JK, Brain K. Barriers to uptake among high-risk individuals declining participation in lung cancer screening: a mixed methods analysis of the UK Lung Cancer Screening (UKLS) trial. BMJ Open. 2015 Jul 14;5(7):e008254. doi: 10.1136/bmjopen-2015-008254. PMID 26173719
- [Background] Lillie SE, Fu SS, Fabbrini AE, Rice KL, Clothier B, Nelson DB, Doro EA, Moughrabieh MA, Partin MR. What factors do patients consider most important in making lung cancer screening decisions? Findings from a demonstration project conducted in the Veterans Health Administration. Lung Cancer. 2017 Feb;104:38-44. doi: 10.1016/j.lungcan.2016.11.021. Epub 2016 Nov 29. PMID 28212998
- [Background] Quaife SL, Marlow LAV, McEwen A, Janes SM, Wardle J. Attitudes towards lung cancer screening in socioeconomically deprived and heavy smoking communities: informing screening communication. Health Expect. 2017 Aug;20(4):563-573. doi: 10.1111/hex.12481. Epub 2016 Jul 11. PMID 27397651
- [Background] Jonnalagadda S, Bergamo C, Lin JJ, Lurslurchachai L, Diefenbach M, Smith C, Nelson JE, Wisnivesky JP. Beliefs and attitudes about lung cancer screening among smokers. Lung Cancer. 2012 Sep;77(3):526-31. doi: 10.1016/j.lungcan.2012.05.095. Epub 2012 Jun 6. PMID 22681870
- [Background] Carter-Harris L, Ceppa DP, Hanna N, Rawl SM. Lung cancer screening: what do long-term smokers know and believe? Health Expect. 2017 Feb;20(1):59-68. doi: 10.1111/hex.12433. Epub 2015 Dec 23. PMID 26701339
- [Background] Roth JA, Carter-Harris L, Brandzel S, Buist DSM, Wernli KJ. A qualitative study exploring patient motivations for screening for lung cancer. PLoS One. 2018 Jul 5;13(7):e0196758. doi: 10.1371/journal.pone.0196758. eCollection 2018. PMID 29975709
- [Background] Triplette M, Kross EK, Mann BA, Elmore JG, Slatore CG, Shahrir S, Romine PE, Frederick PD, Crothers K. An Assessment of Primary Care and Pulmonary Provider Perspectives on Lung Cancer Screening. Ann Am Thorac Soc. 2018 Jan;15(1):69-75. doi: 10.1513/AnnalsATS.201705-392OC. PMID 28933940
- [Background] Kanodra NM, Pope C, Halbert CH, Silvestri GA, Rice LJ, Tanner NT. Primary Care Provider and Patient Perspectives on Lung Cancer Screening. A Qualitative Study. Ann Am Thorac Soc. 2016 Nov;13(11):1977-1982. doi: 10.1513/AnnalsATS.201604-286OC. PMID 27676369
- [Background] Rajupet S, Doshi D, Wisnivesky JP, Lin JJ. Attitudes About Lung Cancer Screening: Primary Care Providers Versus Specialists. Clin Lung Cancer. 2017 Nov;18(6):e417-e423. doi: 10.1016/j.cllc.2017.05.003. Epub 2017 May 10. PMID 28648531
- [Background] Henderson LM, Jones LM, Marsh MW, Brenner AT, Goldstein AO, Benefield TS, Greenwood-Hickman MA, Molina PL, Rivera MP, Reuland DS. Opinions, practice patterns, and perceived barriers to lung cancer screening among attending and resident primary care physicians. Risk Manag Healthc Policy. 2018 Jan 22;10:189-195. doi: 10.2147/RMHP.S143152. eCollection 2017. PMID 29403320
- [Background] Simmons VN, Gray JE, Schabath MB, Wilson LE, Quinn GP. High-risk community and primary care providers knowledge about and barriers to low-dose computed topography lung cancer screening. Lung Cancer. 2017 Apr;106:42-49. doi: 10.1016/j.lungcan.2017.01.012. Epub 2017 Jan 31. PMID 28285693
- [Background] Ersek JL, Eberth JM, McDonnell KK, Strayer SM, Sercy E, Cartmell KB, Friedman DB. Knowledge of, attitudes toward, and use of low-dose computed tomography for lung cancer screening among family physicians. Cancer. 2016 Aug 1;122(15):2324-31. doi: 10.1002/cncr.29944. Epub 2016 Jun 13. PMID 27294476
- [Background] Raz DJ, Wu GX, Consunji M, Nelson RA, Kim H, Sun CL, Sun V, Kim JY. The Effect of Primary Care Physician Knowledge of Lung Cancer Screening Guidelines on Perceptions and Utilization of Low-Dose Computed Tomography. Clin Lung Cancer. 2018 Jan;19(1):51-57. doi: 10.1016/j.cllc.2017.05.013. Epub 2017 Jun 1. PMID 28652090
- [Background] Lewis JA, Petty WJ, Tooze JA, Miller DP, Chiles C, Miller AA, Bellinger C, Weaver KE. Low-Dose CT Lung Cancer Screening Practices and Attitudes among Primary Care Providers at an Academic Medical Center. Cancer Epidemiol Biomarkers Prev. 2015 Apr;24(4):664-70. doi: 10.1158/1055-9965.EPI-14-1241. Epub 2015 Jan 22. PMID 25613118
- [Background] Raz DJ, Wu GX, Consunji M, Nelson R, Sun C, Erhunmwunsee L, Ferrell B, Sun V, Kim JY. Perceptions and Utilization of Lung Cancer Screening Among Primary Care Physicians. J Thorac Oncol. 2016 Nov;11(11):1856-1862. doi: 10.1016/j.jtho.2016.06.010. Epub 2016 Jun 23. PMID 27346412
- [Background] Carter-Harris L, Tan AS, Salloum RG, Young-Wolff KC. Patient-provider discussions about lung cancer screening pre- and post-guidelines: Health Information National Trends Survey (HINTS). Patient Educ Couns. 2016 Nov;99(11):1772-1777. doi: 10.1016/j.pec.2016.05.014. Epub 2016 May 17. PMID 27241830
- [Background] Brenner AT, Malo TL, Margolis M, Elston Lafata J, James S, Vu MB, Reuland DS. Evaluating Shared Decision Making for Lung Cancer Screening. JAMA Intern Med. 2018 Oct 1;178(10):1311-1316. doi: 10.1001/jamainternmed.2018.3054. PMID 30105393
- [Background] Volk RJ, Linder SK, Leal VB, Rabius V, Cinciripini PM, Kamath GR, Munden RF, Bevers TB. Feasibility of a patient decision aid about lung cancer screening with low-dose computed tomography. Prev Med. 2014 May;62:60-3. doi: 10.1016/j.ypmed.2014.02.006. Epub 2014 Feb 8. PMID 24518006
- [Background] Housten AJ, Lowenstein LM, Leal VB, Volk RJ. Responsiveness of a Brief Measure of Lung Cancer Screening Knowledge. J Cancer Educ. 2018 Aug;33(4):842-846. doi: 10.1007/s13187-016-1153-8. PMID 27966194
- [Background] Bellinger C, Pinsky P, Foley K, Case D, Dharod A, Miller D. Lung Cancer Screening Benefits and Harms Stratified by Patient Risk: Information to Improve Patient Decision Aids. Ann Am Thorac Soc. 2019 Apr;16(4):512-514. doi: 10.1513/AnnalsATS.201810-690RL. No abstract available. PMID 30620619
- [Background] Dharod A, Bellinger C, Foley K, Case LD, Miller D. The Reach and Feasibility of an Interactive Lung Cancer Screening Decision Aid Delivered by Patient Portal. Appl Clin Inform. 2019 Jan;10(1):19-27. doi: 10.1055/s-0038-1676807. Epub 2019 Jan 9. PMID 30625501
- [Background] Miller DP Jr, Weaver KE, Case LD, Babcock D, Lawler D, Denizard-Thompson N, Pignone MP, Spangler JG. Usability of a Novel Mobile Health iPad App by Vulnerable Populations. JMIR Mhealth Uhealth. 2017 Apr 11;5(4):e43. doi: 10.2196/mhealth.7268. PMID 28400354
- [Background] Katki HA, Kovalchik SA, Petito LC, Cheung LC, Jacobs E, Jemal A, Berg CD, Chaturvedi AK. Implications of Nine Risk Prediction Models for Selecting Ever-Smokers for Computed Tomography Lung Cancer Screening. Ann Intern Med. 2018 Jul 3;169(1):10-19. doi: 10.7326/M17-2701. Epub 2018 May 15. PMID 29800127
- [Background] Pinsky PF, Bellinger CR, Miller DP Jr. False-positive screens and lung cancer risk in the National Lung Screening Trial: Implications for shared decision-making. J Med Screen. 2018 Jun;25(2):110-112. doi: 10.1177/0969141317727771. Epub 2017 Sep 20. PMID 28929865
- [Background] Fagerlin A, Zikmund-Fisher BJ, Ubel PA. Helping patients decide: ten steps to better risk communication. J Natl Cancer Inst. 2011 Oct 5;103(19):1436-43. doi: 10.1093/jnci/djr318. Epub 2011 Sep 19. PMID 21931068
- [Background] Hawley ST, Zikmund-Fisher B, Ubel P, Jancovic A, Lucas T, Fagerlin A. The impact of the format of graphical presentation on health-related knowledge and treatment choices. Patient Educ Couns. 2008 Dec;73(3):448-55. doi: 10.1016/j.pec.2008.07.023. Epub 2008 Aug 27. PMID 18755566
- [Background] Hoffman AS, Hempstead AP, Housten AJ, Richards VF, Lowenstein LM, Leal VB, Volk RJ. Using a Patient Decision Aid Video to Assess Current and Former Smokers' Values About the Harms and Benefits of Lung Cancer Screening With Low-Dose Computed Tomography. MDM Policy Pract. 2018 Apr 19;3(1):2381468318769886. doi: 10.1177/2381468318769886. eCollection 2018 Jan-Jun. PMID 30288444
- [Background] Pignone MP, Howard K, Brenner AT, Crutchfield TM, Hawley ST, Lewis CL, Sheridan SL. Comparing 3 techniques for eliciting patient values for decision making about prostate-specific antigen screening: a randomized controlled trial. JAMA Intern Med. 2013 Mar 11;173(5):362-8. doi: 10.1001/jamainternmed.2013.2651. PMID 23400279
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Lowenstein LM, Richards VF, Leal VB, Housten AJ, Bevers TB, Cantor SB, Cinciripini PM, Cofta-Woerpel LM, Escoto KH, Godoy MC, Linder SK, Munden RF, Volk RJ. A brief measure of Smokers' knowledge of lung cancer screening with low-dose computed tomography. Prev Med Rep. 2016 Jul 26;4:351-6. doi: 10.1016/j.pmedr.2016.07.008. eCollection 2016 Dec. PMID 27512650
- [Background] Bangor A, Kortum PT, Miller JT. An Empirical Evaluation of the System Usability Scale. Int J Human-Computer Interact. 2008;24(6):574-594. doi:10.1080/10447310802205776
- [Background] Henderson LM, Marsh MW, Benefield TS, Jones LM, Reuland DS, Brenner AT, Goldstein AO, Molina PL, Maygarden SJ, Rivera MP. Opinions and Practices of Lung Cancer Screening by Physician Specialty. N C Med J. 2019 Jan-Feb;80(1):19-26. doi: 10.18043/ncm.80.1.19. PMID 30622199
- [Derived] Miller DP, Snavely AC, Dharod A, Brenner AT, Wright E, Stradtman L, Bellinger CR, Bundy R, Volk RJ, Hamburger E, Ferrari RM, Randazzo A, Reuland DS. A Direct-to-Patient Digital Health Program for Lung Cancer Screening: A Randomized Clinical Trial. JAMA. 2025 Nov 25;334(20):1807-1815. doi: 10.1001/jama.2025.17281. PMID 41114973

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants are considered enrolled in this study when they are randomly selected by the study team to receive an invitation to use mPATH. Of the 26,909 people who were sent invitation messages, 3,267 visited the mPATH program and completed eligibility questions, and 1,333 were confirmed eligible for LCS and subsequently randomized.
Groups:
- Primary Care Providers: Primary care providers who completed a survey about their experiences.
Period: Overall Study
Arm/Group | mPATH-Lung | Usual Care (CONTROL) | Primary Care Providers
Started | 669 | 664 | 89
Completed | 669 | 664 | 89
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were determined to be eligible for LCS based on their responses to initial questions in the mPATH program were randomized into either the intervention or enhanced usual care arm. No baseline characteristics were collected for participants in the "Primary Care Providers" arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | mPATH-Lung | Usual Care (CONTROL) | Total
Number analyzed (Participants) | 669 | 664 | 1333
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 458 | 483 | 941
  >=65 years | 211 | 181 | 392
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 425 | 439 | 864
  Male | 244 | 225 | 469
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 13 | 18
  Not Hispanic or Latino | 664 | 651 | 1315
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 114 | 118 | 232
  White | 533 | 521 | 1054
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 22 | 25 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Electronic Health Record-verified Completion of a Chest CT Scan
Description: Participants who have completed any chest CT within 16 weeks of study randomization, as determined by electronic health record review
Time Frame: Within 16 weeks of enrollment
Population: This population includes all participants who used the mPATH program to the point of randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | mPATH-Lung | Usual Care (CONTROL)
Number analyzed (Participants) | 669 | 664
Participants | 164 | 113

2. Secondary Outcome: LCS Screening Decision
Description: Patient intention to receive LCS as measured by a survey item in the mPATH-Lung group only
Time Frame: Up to 16 weeks after day of enrollment
Reporting Status: Not Posted

3. Secondary Outcome: Proportion of Patients With LCS Clinic Visits Scheduled
Description: The proportion of patients in each arm who have scheduled a LCS clinic visit, whether or not the visit is completed
Time Frame: 16 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Proportion of Patients With LCS Clinic Visits Completed
Description: The proportion of patients in each arm who have completed a LCS clinic visit
Time Frame: 16 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Proportion of Patients With LCS Scans Ordered
Description: The proportion of patients in each arm for whom a LCS scan was ordered
Time Frame: 16 weeks
Reporting Status: Not Posted

6. Secondary Outcome: LCS Clinic Referral Requested Through mPATH
Description: The proportion of patients in mPATH-Lung arm who completed a referral form with request for appointment.
Time Frame: 16 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Lung Cancer Screening Test Results
Description: The results of a completed lung cancer screening CT, reported using the Lung-RADS classification
Time Frame: 16 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Number of LCS False Positives
Description: A Lung-RADS 3 or 4 result with a negative completed work-up for lung cancer or no diagnosis of lung cancer within 12 months of the scan.
Time Frame: 1 year
Reporting Status: Not Posted

9. Secondary Outcome: Invasive Procedures Following LCS Scan
Description: The proportion of patients in each arm who undergo an invasive procedure following a LCS scan
Time Frame: 1 year
Reporting Status: Not Posted

10. Secondary Outcome: Proportion of Patients With Complications Following LCS
Description: The proportion of patients in each arm who experience a complication from an invasive procedure following a LCS scan
Time Frame: 1 year
Reporting Status: Not Posted

11. Secondary Outcome: Number of Diagnosed Lung Cancers
Description: Number of diagnosed lung cancers (detected by screening or other) within 16 months of randomization
Time Frame: 16 months after randomization
Reporting Status: Not Posted

12. Secondary Outcome: How Diagnosed Lung Cancers Were Detected
Description: Proportion of patients who had lung cancers detected related to screening or incidentally.
Time Frame: 16 months after randomization
Reporting Status: Not Posted

13. Secondary Outcome: Stage of Lung Cancers Diagnosed
Description: Stage of lung cancers diagnosed
Time Frame: 16 months after randomization
Reporting Status: Not Posted

14. Secondary Outcome: Overscreening
Description: The proportion of patients with screen diagnosed lung cancer who are deemed too ill for potentially curative surgery by blinded chart review.
Time Frame: 1 year
Reporting Status: Not Posted

15. Secondary Outcome: Reach of Digital Outreach Strategy
Description: The proportion of patients sent a digital invitation who complete the eligibility questions on the study website.
Time Frame: 16 weeks
Population: All individuals who were sent an invitation to use the mPATH program.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants Invited to Use mPATH: All individuals who were sent an invitation to use the mPATH program.
Arm/Group | All Participants Invited to Use mPATH
Number analyzed (Participants) | 26909
Participants | 3267

16. Secondary Outcome: Completion of mPATH-Lung Program
Description: The proportion of patients randomized to mPATH-Lung who complete the mPATH-Lung program to the point of indicating their screening decision.
Time Frame: 16 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Description: No adverse event details were collected for participants in the "Primary Care Providers" arm.
Arm/Group | mPATH-Lung | Usual Care (CONTROL)
All-Cause Mortality (participants affected / at risk) | 0/669 | 0/664
Serious Adverse Events (participants affected / at risk) | 0/669 | 0/664
Other Adverse Events (participants affected / at risk) | 0/669 | 0/664

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT04083859/Prot_SAP_002.pdf
  • Informed Consent Form (2023-11-28): https://cdn.clinicaltrials.gov/large-docs/59/NCT04083859/ICF_003.pdf